CLINICAL TRIAL: NCT06010914
Title: Drug Use Investigation of Darolutamide in Addition to Standard Androgen Deprivation Therapy (ADT) and Docetaxel in Patients With Metastatic Hormone-sensitive Prostate Cancer (mHSPC)
Brief Title: A Study to Learn More About How Safe Darolutamide is Under Real-world Conditions in Participants With Metastatic Hormone-Sensitive Prostate Cancer
Acronym: DADOX
Status: Active, not recruiting | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 22523
Record Dates: First submitted 2023-08-21; First posted 2023-08-25 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Hormone-sensitive Prostate Cancer (mHSPC)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- mHSPC patients to treat with darolutamide in combination with docetaxel and ADT: Patients over the age of 18 years with a diagnosis of mHSPC and for whom a decision to treat with darolutamide in combination with docetaxel and ADT has been made by the treating physician before study enrollment.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — Following the manner of observational study, no intervention will be provided in the study.
  The decision on the dose and duration of treatment is solely at the discretion of the treating physician, based on the recommendations written in the local product information.

SUMMARY:
This is an observational study in which only data are collected from participants receiving their usual treatment.

In this study, data will be collected and studied from men with metastatic hormone-sensitive prostate cancer (mHSPC). Prostate cancer is a common cancer in men that starts in the prostate gland, a male reproductive gland found below the bladder. Metastatic means that the cancer has spread to other parts of the body. Hormone-sensitive means it can be treated with hormone-therapy such as androgen deprivation therapy (ADT). ADT lowers the level of testosterone, a male hormone, and slows down the growth of cancer cells.

Men with mHSPC and who have been decided by their own doctors to be treated with darolutamide in combination with ADT and docetaxel can join this study. Darolutamide works by blocking the testosterone signals to slow the growth of the cancer cells. Docetaxel is a medicine used to treat different types of cancer. It works by stopping the growth and spread of cancer cells.

Darolutamide in combination with docetaxel and ADT is an approved treatment for men with mHSPC. It was approved based on a study called ARASENS. More information is needed on how safe darolutamide is when given with ADT and docetaxel in Japanese men with mHSPC.

The main purpose of this study is to collect information about the safety of this combination treatment in Japanese participants with mHSPC under real-world conditions.

The main information that researchers will collect:

Number and severity of heart-related medical problems participants have during the treatment

Other information that researchers will collect:

Number and severity of all medical problems participants have during the study

Age and other information about the participants such as their illness, medical history, and other medicines taken at the same time

Treatment pattern of darolutamide such as the amount of medicine given, the duration for which it is given, and any changes made to the treatment

Data will be collected from August 2023 to July 2026. Researchers will observe participants from the start of darolutamide treatment until 30 days after they receive their last dose of docetaxel, which is expected to be approximately 6 months for each participant.

In this study, data from regular health visits will be collected. No visits or tests are required as part of this study.

ELIGIBILITY:
Inclusion Criteria:

* Men over the age of 18 years
* Histologically or cytologically confirmed adenocarcinoma prostate cancer
* Metastatic disease confirmed either by a positive bone scan, or for soft tissue or visceral metastases, either by contrast-enhanced abdominal/pelvic/chest computed tomography (CT) or magnetic resonance imaging (MRI) scan
* Patients diagnosed with mHSPC by the investigator under routine clinical practice, and must be judged appropriate for/decided to be treated with darolutamide plus ADT and docetaxel therapy by the investigator under routine clinical practice
* ADT (GnRH agonist/antagonist or orchiectomy) before or simultaneous treatment with darolutamide
* Signed informed consent

Exclusion Criteria:

* Participation in an investigational program with interventions outside of routine clinical practice
* Contraindications according to the local marketing authorization
* Previous treatment with darolutamide

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male patients with a diagnosis of mHSPC will be enrolled after the decision for treatment with darolutamide in combination with docetaxel and ADT has been made by the physician or a delegate.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-10-09 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with cardiac treatment-emergent adverse events (TEAEs) | From the start of darolutamide treatment to 30 days after the last dose of docetaxel
  Incidence of cardiac disorders (TEAEs based on MedDRA SOC), including severity, seriousness, onset date and outcome.
Outcomes of cardiac TEAEs | From the start of darolutamide treatment to 30 days after the last dose of docetaxel
  Causal relationship (i.e. if a specific AE is related to daroluatmide) between darolutamide and cardiac disorders.
Dose modifications due to cardiac TEAEs | From the start of darolutamide treatment to 30 days after the last dose of docetaxel
  Action taken related to darolutamide (dose modifications and time periods).

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) | From the start of darolutamide treatment to 30 days after the last dose of docetaxel
  Occurrence of AEs, including severity, seriousness, onset date and outcome. Adverse event (AE): Any untoward medical occurrence in a patient administered a pharmaceutical product and which does not necessarily have to have a causal relationship (association) with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of the product, whether or not related to the product.
Patient demographics/characteristics | From the start of darolutamide treatment to 30 days after the last dose of docetaxel
  All background data such as patient demographics, diagnosis and prior treatment, past medical history, concomitant diseases, and concomitant medications.
  * Baseline characteristics (vital signs, Gleason Score, ECOG PS, PSA)
  * Prostate cancer history
  * Prior and ongoing Co-morbidities
  * Darolutamide, GnRH agonist/antagonist, docetaxel use:
    * Initiation and termination dates and reasons for ending treatment.
Descriptive summary of dosing patterns of darolutamide | From the start of darolutamide treatment to 30 days after the last dose of docetaxel
Outcomes of AEs | From the start of darolutamide treatment to 30 days after the last dose of docetaxel
  Causal relationship (i.e. if a specific AE is related to daroluatmide) between darolutamide and AE/ADR, and action taken related to darolutamide (dose modifications and time periods).
Dose modifications due to AEs | From the start of darolutamide treatment to 30 days after the last dose of docetaxel
  Dosing patterns.

CONTACTS AND LOCATIONS:
Locations (1):
- Many Locations, Multiple Locations, Japan

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.